CLINICAL TRIAL: NCT04908332
Title: Effect of a Nursing Intervention on the Mother-baby Kangaroo Interaction at Home in Bogotá
Brief Title: Effect of Kangaroo Baby Massage on Mother-infant Interaction at Home
Acronym: KBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Nubia Castiblanco Lopez, student Nursing PhD, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNColombia KBM
Record Dates: First submitted 2021-05-18; First posted 2021-06-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-05

CONDITIONS: Premature; Low Birth Weight; Mother-Infant Interaction; Gain, Weight; Depression, Post-Partum; Breastfeeding; Feeding, Breast
Keywords: Massage; Kangaroo mother care; low birth weight infant; premature infant; Mother- infant interaction; domiciliary; Nursing; home health nursing; telenursing
MeSH Terms: conditions — Premature Birth; Weight Gain; Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Two interventions groups of 34 each, participated in the study. The first group received Nursing intervention Kangaroo Baby Massage KBM at home and the second group received Kangaroo position KP at home, the KBM will start when the infant arrives at home until they leave the kangaroo position. The KP will measure since the baby arrive at home until leave the kangaroo position.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The infant-mother dyads will not be Know that there are two different interventions in each group. This leads to greater adherence to treatment.
  The researchers: there will be two research assistants who will receive capacity regardless of the group of participants they are going to train, the main researcher will not carry out the training to the mothers and will be blinded.
  The nursing assistant in charge of weighing the baby and the pediatrician who determines the time of the kangaroo position. They will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo baby Massage (Experimental): The mother will apply the massage. The baby kangaroo will be exposed to the KBM for 10 minutes once a day during the time that the infant need to stay in kangaroo position at home. If the baby wakes up and wants to eat the KBM will be interrupted immediately and the baby will be fed, The temperature will be measured before and after the intervention. The massage will begin 60 minutes after the feed.
  Interventions: Behavioral: Kangaroo Baby Massage
- Kangaroo position (Active Comparator): The infant must be in Kangaroo position with the mother semi sitting on bed with elevation of at least 30 degrees during 10 minutes every day until the infant doesn´t need to stay in kangaroo position at home.The temperature will be measured 60 minutes after the feed and 10 minutes after KP. If the baby wakes up and wants to eat the KP will be interrupted immediately and the baby will be fed, then the KP will be completed of time ( 10 minutes) to measure the temperature.
  Interventions: Behavioral: Kangaroo Baby Massage

INTERVENTIONS:
Behavioral: Kangaroo Baby Massage — The Kangaroo Baby Massage is an intervention that arose from nursing practice in 1996. It is a therapy that does not require an incubator, fuses massage, kangaroo position and music. KBM is available on video
  Other Names: Masaje al Bebé Canguro; Nursing intervention KBM

SUMMARY:
The objective of this randomized clinical trial will determine the effectiveness of nursing intervention (Kangaroo Baby Massage) on the interaction between mothers and premature, low birth weight infants at home The dyad mother- infant of the control group will receive Kangaroo position KP and the dyad mother- infant mothers of the intervention group will receive the Kangaroo Baby Massage KBM

DETAILED DESCRIPTION:
Participants and methods: 68 dyads mother-infant will randomize, 34 in intervention KBM group and 34 in control group KP, previous they meet inclusion criteria and accept their participation through informed consent. weight gain and Kangaroo position days at home will be the primaries outcomes. The Alert states, Types of BC feeding, Perceived maternal parental self-efficacy and Postnatal depression. Will be secondary outcomes.

Barnard's mother-child interaction theory supports the study

ELIGIBILITY:
Inclusion Criteria

* Prematures and low birth weight infants in Kangaroo position with a chronological age less than 3 months
* The mothers take care the infant at home
* Baby with a weight equal to or greater than 1800 grams at the time of entry to the study.
* Baby whose birth was institutional or extra-institutional.
* Mothers with training in the Kangaroo Mother Program
* Children controlled in the Ambulatory Kangaroo Mother Program

Exclusion Criteria

* Children diagnosed with intraventricular hemorrhages grade III and IV or congenital malformations
* Children who have more than one ambulatory kangaroo control
* Children who have been at home for more than 3 days without starting the ambulatory kangaroo control
* Babies with infections and other pathologies that require hospitalization during the study
* Presence of infectious diseases and other pathologies in the mother that require hospitalization
* Mother confirmed with positive test for covid 19 at the moment of the randomization
* Mothers with cognitive problems or mental disorders.

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
weight | Through study completion, an average of 20 days
  Weight gain after randomization up to infant doesn´t need to stay in kangaroo position at home.
Kangaroo position days at home | Through study completion, an average of 20 days
  Number days that the infant needs to stay in kangaroo position at home

SECONDARY OUTCOMES:
Alert states | Through study completion, an average of 20 days
  The mother will observe and record YES OR NO the baby woke up during the intervention
Types of feeding | Through study completion, an average of 20 days
  The mother will report whether or not the baby fed during the intervention and will identify the type of feeding (exclusive breast milk, formula or mixed)
Perceived maternal parental self-efficacy | Given by a self-report provided by the mother of the perceived maternal parental self-efficacy questionnaire on day 1 before randomization and day 7 and 14 after randomization
  The questionnaire contains 20 items with a Likert scale (1. Totally disagree, 2. disagree, 3. agree and 4. totally agree) the minimum value is 20 and the maximum is 80 and the higher scores means a better outcome.
Postnatal depression | Given by a self-report provided by the mother of the Edinburgh Postnatal Depression Scale on day 1 before randomization and day 7 and 14 after randomization
  . This scale contains 10 points of 0, 1, 2 and 3 are given according to the increase in the severity of the symptom. The points for questions 3, 5, 6, 7, 8, 9, 10 are scored in reverse order (3, 2, 1, 0). All points are added together to give the total score. A score of 10+ means worse outcome and shows the probability of depression

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Vesga Gualdron, Professor, Study Director — Universidad Nacional de Colombia; Fred Manrique Abril, Professor, Study Director — Universidad Nacional de Colombia; Nubia Castiblanco Lopez, PhD student, Principal Investigator — Universidad Nacional de Colombia
Locations (1):
- Programa canguro ambulatorio, Bogotá, Colombia

REFERENCES:
- [Background] Chan GJ, Labar AS, Wall S, Atun R. Kangaroo mother care: a systematic review of barriers and enablers. Bull World Health Organ. 2016 Feb 1;94(2):130-141J. doi: 10.2471/BLT.15.157818. Epub 2015 Dec 3. PMID 26908962
- [Background] Premji SS, Currie G, Reilly S, Dosani A, Oliver LM, Lodha AK, Young M. A qualitative study: Mothers of late preterm infants relate their experiences of community-based care. PLoS One. 2017 Mar 23;12(3):e0174419. doi: 10.1371/journal.pone.0174419. eCollection 2017. PMID 28334033
- [Background] Rangey PS, Sheth M. Comparative Effect of Massage Therapy versus Kangaroo Mother Care on Body Weight and Length of Hospital Stay in Low Birth Weight Preterm Infants. Int J Pediatr. 2014;2014:434060. doi: 10.1155/2014/434060. Epub 2014 May 25. PMID 24976830
- [Background] Holditch-Davis D, White-Traut R, Levy J, Williams KL, Ryan D, Vonderheid S. Maternal satisfaction with administering infant interventions in the neonatal intensive care unit. J Obstet Gynecol Neonatal Nurs. 2013 Nov-Dec;42(6):641-54. doi: 10.1111/1552-6909.12255. PMID 25803213
- [Background] Pados BF, McGlothen-Bell K. Benefits of Infant Massage for Infants and Parents in the NICU. Nurs Womens Health. 2019 Jun;23(3):265-271. doi: 10.1016/j.nwh.2019.03.004. Epub 2019 May 3. PMID 31059673
- [Background] Vargas-Porras C, Roa-Diaz ZM, Barnes C, Adamson-Macedo EN, Ferre-Grau C, De Molina-Fernandez MI. Psychometric Properties of the Spanish Version of the Perceived Maternal Parenting Self-efficacy (PMP S-E) Tool for Primiparous Women. Matern Child Health J. 2020 May;24(5):537-545. doi: 10.1007/s10995-019-02860-y. PMID 31916144
- [Background] Stuebe A. Should Infants Be Separated from Mothers with COVID-19? First, Do No Harm. Breastfeed Med. 2020 May;15(5):351-352. doi: 10.1089/bfm.2020.29153.ams. Epub 2020 Apr 9. No abstract available. PMID 32271625